CLINICAL TRIAL: NCT02541045
Title: Clinical Trial to Evaluate the Efficacy of Metadoxine as a Therapy for Patients With Non-alcoholic Steatohepatitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of resources to finance the project
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, MARIA DE FATIMA HIGUERA DE LA TIJERA, MD, MSc., Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DI/15/108/03/48
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: non-alcoholic steatohepatitis; metadoxine; efficacy; therapy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — metadoxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Placebo (Placebo Comparator): Placebo
  Interventions: Other: placebo
- Group 2: Metadoxine (Experimental): therapy with metadoxine
  Interventions: Drug: metadoxine

INTERVENTIONS:
Drug: metadoxine — metadoxine 500mg tablets: 1 Tablet by mouth twice in day during 6 months
  Other Names: Abrixone, Metadoxil
  Arms: Group 2: Metadoxine
Other: placebo — placebo tablets: 1 Tablet by mouth twice in day during 6 months
  Arms: Group 1: Placebo

SUMMARY:
The aim of this study is to evaluate the efficacy of metadoxine as a therapy for patients with biopsy-proven non-alcoholic steatohepatitis.

DETAILED DESCRIPTION:
Type and design of the study: A randomized, placebo-controlled, double-blind, clinical trial to evaluate the efficacy of metadoxine as a therapy in patients with biopsy-proven nonalcoholic steatohepatitis.

Population: Non-diabetic patients with nonalcoholic steatohepatitis diagnosed by liver biopsy through the "nonalcoholic fatty liver disease activity score" (NAS)> 3.

Sample size: Considering a difference of at least 30% between groups, a confidence level of 95% (two-sided, significance 0.05), a statistical power of 80%, and an additional 20% for possible losses, we need 54 patients per group.

Variables:

Independent: Treatment group (metadoxine / placebo).

Dependents:

* "Nonalcoholic fatty liver disease activity score" (NAS):0 a 8
* Degree of liver steatosis: 0 a 3
* Degree of lobular inflammation: 0 a 3
* Degree of ballooning: 0 a 2
* Degree of fibrosis: 0 a 2
* Weight: Kg
* Body mass index: Kg/m2
* Waist circumference: cm
* Serum alanine aminotransferase: U/L
* Serum aspartate aminotransferase: U/L

Methods:

Those meeting the selection criteria will be invited to participate in this study, those who agree to participate must sign the consent form and will be randomized to placebo or metadoxine group. The duration of the therapy will be 6 months and after this period a second liver biopsy will be performed to assessed the improvement on liver histology.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic patients,
* Overweight or with obesity degrees I, II or III according to WHO criteria (BMI ≥ 25),
* With evidence of liver steatosis in the ultrasonography,
* With biopsy-proven nonalcoholic steatohepatitis, with ≥ 3 in the NAS score (at least 1 point for liver steatosis, at least 1 point for lobular inflammation, and at least 1 point for ballooning),
* With or without fibrosis in the liver biopsy, but if it is present must be ≤ 2 on a scale of 4, where 4 is equivalent to cirrhosis.

Exclusion Criteria:

* Cirrhosis,
* Diabetes,
* Heavy alcohol intake ( ≥ 20 g / day), ≥ 8 points in the "Alcohol Use Disorders Identification Test" (AUDIT),
* Acute or chronic hepatitis C,
* Acute or chronic hepatitis B,
* Immunodeficiency acquired syndrome
* Pregnant women,
* In the last year, history of herbal consumption, total parenteral nutrition, amiodarone, methotrexate, hormonal contraceptives, steroids, tamoxifen, valproic acid or any other drug associated with the development of liver steatosis.
* Uncontrolled hypothyroidism or hyperthyroidism,
* Any uncontrolled chronic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2024-03 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
improvement in the degree of non-alcoholic fatty liver disease score (NAS) | 6 months
  Non-alcoholic fatty liver disease score (NAS) is an histological classification to assessed the severity of liver steatosis, lobular inflammation and ballooning in the liver biopsy. It is measured on a scale from 0 to 8

SECONDARY OUTCOMES:
improvement in liver steatosis measured on a scale from 0 to 3 | 6 months
  Liver biopsy: measured on a scale from 0 to 3
improvement in lobular inflammation measured on a scale from 0 to 3 | 6 months
  Liver biopsy: measured on a scale from 0 to 3
improvement in ballooning measured on a scale from 0 to 2 | 6 months
  Liver biopsy: measured on a scale from 0 to 2
improvement in alanine aminotransferase serum levels | 6 months
improvement in aspartate aminotransferase serum levels | 6 months
improvement in the degree of liver fibrosis measured on a scale from 0 to 2 | 6 months
  Liver biopsy: measured on a scale from 0 to 2
to compare the occurrence of adverse effects between groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Higuera-de la Tijera, MD, MSc., Study Director — Hospital General de México
Locations (1):
- Hospital General de México, Mexico City, Mexico City, Mexico